CLINICAL TRIAL: NCT07347600
Title: A Prospective Non-interventional Study to Evaluate the Effectiveness and Safety of Inavolisib in Patients With Endocrine-resistant, PIK3CA-mutated, Hormone Receptor-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer (reaINAVO)
Brief Title: A Study to Evaluate the Effectiveness and Safety of Inavolisib in Participants With Endocrine-resistant, PIK3CA-mutated, Hormone Receptor-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer
Acronym: reaINAVO
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML46361
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; palbociclib; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inavolisib: Participants with endocrine-resistant, PIK3CA-mutated, HR+, HER2-, LA/mBC, following on or after completing adjuvant endocrine therapy will be observed for effectiveness and safety of inavolisib.
  Interventions: Drug: Inavolisib; Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Inavolisib — Inavolisib will be administered at the discretion of the physician in accordance with local clinical practice and local labeling.
  Other Names: GDC-0077
Drug: Palbociclib — Palbociclib will be administered at the discretion of the physician in accordance with local clinical practice and local labeling.
Drug: Fulvestrant — Fulvestrant will be administered at the discretion of the physician in accordance with local clinical practice and local labeling.

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of inavolisib based regimen in participants with endocrine-resistant, phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha gene (PIK3CA)-mutated, hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) locally advanced or metastatic breast cancer (LA/mBC), following on or after completing adjuvant endocrine therapy in routine clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with endocrine-resistant, PIK3CA-mutated, HR+/HER2- LA/mBC, following recurrence on or after completing adjuvant endocrine therapy
* Participants must receive the treatment of inavolisib for the first time
* PIK3CA mutation status should be detected by a National Medical Products Administration (NMPA)-approved or validated assay [Polymerase Chain Reaction (PCR) or Next Generation Sequencing (NGS)] by testing of blood or tumor tissue prior to the initiation of inavolisib

Exclusion Criteria:

* Participants for which the treatment with inavolisib is not indicated per prescribing information. If the participant starts palbociclib and fulvestrant first, and starts inavolisib after getting a PIK3CA mutation-positive test result later, the palbociclib and fulvestrant will not be deemed as a different line of therapy. However, the medical order of PIK3CA mutation test must be made before or at the same time with the prescription of palbociclib and fulvestrant
* Participants not receiving treatment for LA/mBC with inavolisib according to standard of care (SOC) and in line with the current summary of product characteristics (SPC)/local labeling
* At the investigator's discretion, any reason that makes the participant hard to follow up or unsuitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with endocrine-resistant, PIK3CA-mutated, HR+, HER2-, LA/mBC, following on or after completing adjuvant endocrine therapy in routine clinical practice in China.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-09-09 (Estimated)

PRIMARY OUTCOMES:
Real-world Progression-free Survival (rwPFS) | From index date (date of first prescription of inavolisib) to first occurrence of disease progression (PD)/death from any cause (up to approximately 36 months)

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately 36 months
Real-world Time to Progression (rwTTP) | From index date to first occurrence of PD (up to approximately 36 months)
Number of Participants With Real-world Tumor Response (rwTR) to the Treatment | Up to approximately 36 months
Real-world Duration of Response (rwDoR) | From onset of first tumor response to first occurrence of PD or death from any cause (up to approximately 36 months)
Real-world Time-to-treatment Discontinuation (rwTTD) | From index date to inavolisib discontinuation, new anti-cancer therapy initiation or death from any cause (up to approximately 36 months)
Real-world Time to Next Treatment (rwTTNT) | From index date to new anti-cancer therapy (up to approximately 36 months)
Real-world Time to Chemotherapy (rwTTC) | From index date to date of chemotherapy initiation (up to approximately 36 months)
Treatment Duration of Inavolisib | Up to approximately 36 months
Total Dose of Inavolisib Received | Up to approximately 36 months
Number of Participants Who Experience Dose Modification, Including Missing Doses, Dose Interruption, Dose Reduction, or Early Discontinuation | Up to approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No